CLINICAL TRIAL: NCT02665143
Title: A Phase I-II Randomized Trial of a Combination of Nintedanib/Placebo in Combination With Induction Chemotherapy for Patients With Refractory or First Relapse Acute Myeloid Leukemia
Brief Title: A Randomized Trial of a Combination of Nintedanib/Placebo in Combination With Induction Chemotherapy for Patients With Refractory or First Relapse Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1507016193
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
Keywords: acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nintedanib and AML induction (Experimental): The AML induction regimen combines Idarubicin 12mg/m2/d day 1 to 3 and Cytarabine 0.667g/m2/d CIV day 1 to 3. Based on the phase I dose, in the randomized phase II, the combination will be compared with chemotherapy+placebo. Nintedanib or placebo will be added at day 8 and continued until end of cycle .
  Interventions: Drug: Nintedanib and AML induction

INTERVENTIONS:
Drug: Nintedanib and AML induction — The AML induction regimen combines Idarubicin 12mg/m2/d day 1 to 3 and Cytarabine 0.667g/m2/d CIV day 1 to 3. In the phase I part, all patients will receive the combination with Nintedanib 200mg bid begun at day 8 and continued until end of cycle. If a significant incidence of dose limiting toxicities is demonstrated, Nintedanib will be given at a lower dose level (150mg bid).
  Other Names: Phase II Open Label

SUMMARY:
The purpose of this study is to determine if a combination of nintedanib+ induction chemotherapy can be an effective strategy for patients where outcome of relapse/refractory acute myeloid leukemia (AML) is poor.

DETAILED DESCRIPTION:
This study will conducted as a Phase 1/Phase 2 trial.

The primary objective of Phase 1 is to determine the safety and tolerability of a combination of Nintedanib + induction chemotherapy in patients with acute myeloid leukemia.

The primary objective of Phase 2 is to determine the efficacy (rate of CR/CRp/CRi) of Nintedanib+ induction vs Placebo+ induction.

The secondary objectives of this study include: determining the overall response rate according to IWG AML 2003 criteria, the toxicity profile and safety of the combination, the percentage of patients bridging to transplantation, the overall survival, leukemia free survival including analysis with censoring at HSCT and rates of haematological improvement according to IWG MDS 2006 criteria. In addition, exploratory correlative studies will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML according to WHO 2008 criteria. Therapy related AML may be included if off treatment for their prior malignancy for more than 2 years and in complete remission. AML arising after documented MPD is excluded.
* Patient must meet one of the following criteria: a/ patient refractory to one or two standard induction regimens b/ patients with a first untreated relapse within 2 years of documentation of complete remission. Patients relapsing after allogeneic stem cell transplantation are eligible if more than 6 months after transplantation and without signs of active GVHD.
* Patient may have been pre treated with intermediate to high dose cytarabine if the day of the last infusion was at least 90 days before the inclusion.
* ECOG performance status of 2 or less
* Patient is willing to participate to the study, has the ability to adhere to the study visit schedule and other protocol procedures, and has the ability to understand and sign an inform consent form.
* Women of childbearing potential must agree to use effective contraception without interruption throughout the study and for 3 months after the end of treatment;
* Men must agree to not conceive during the treatment and to use effective contraception during the treatment period (including periods of dose reduction or temporary suspension) and for 3 months after the end of treatment if their partner is of childbearing potential.

Exclusion Criteria:

* Patient with documented acute promyelocytic leukemia and/or PML-RAR transcript.
* Patient relapsing more than 2 years after initial remission.
* Use of any active treatment for relapse including but not restricted to chemotherapy, targeted agents, hypomethylating agents or investigational drugs. Use of hydroxyurea up to 6g per day for cytoreduction is allowed for a maximum of 30 days prior treatment.
* Patients with clinical evidence of active CNS disease at enrollment
* LVEF below 45% or lifetime exposure to anthracyclines over 350mg/m2 of daunorubicin equivalent
* Liver function tests: ASAT ALAT above 2.5 ULN, total bilirubin above 2.5 ULN in the absence of Hemolysis or diagnosis of Gilbert's syndrome
* Serum creatinine above 2.0mg/dl
* Any sign of active uncontrolled disease including but not restricted to cardiac disease, infections, hepatitis. Any severe chronic disease potentially interfering with the protocol including HIV infection, active hepatitis B or C. It includes major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
* Documented platelet refractoriness
* Patient has a history of GI surgery, procedures or conditions that might interfere with the absorption or swallowing of the study drugs .
* Women who are or pregnant, or who are currently breastfeeding
* Prior treatment with nintedanib or any other VEGFR inhibitor
* Known hypersensitivity to nintedanib, any other trial drug, or their excipients
* Persistence of any clinically relevant (CTCAE grade 2 or above) non-hematological toxicities from previous AML therapy
* Active alcohol or drug abuse
* Any other condition that, according to the investigator, may forbid the administration of the idarubicin+cytarabine regimen
* Therapeutic anticoagulation with INR modifying drug of or use of antiplatelet therapy (with the exception of low dose aspirin<325mg/d)
* Any other malignancies requiring an active treatment within the past year other than basal cell skin cancer or carcinoma in situ of the cervix. Patients actively treated with hormonotherapy for prostate cancer or breast cancer are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Prebet, MD,PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Nintedanib and AML Induction
Started | 6
Completed | 6
Not Completed | 0
Period: Phase 2
Arm/Group | Nintedanib and AML Induction
Started | 19 (19 Participants were enrolled in Phase 2.)
Completed 0 Cycles | 1
Completed 1 Cycle | 12
Completed 2 Cycles | 3
Completed 3 Cycles | 3
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 6 Phase 1 patients and 19 Phase 2 patients.
Arm/Group | Nintedanib and AML Induction
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: There were 6 Phase 1 patients and 19 Phase 2 patients.
  Participants
    Phase 1: number analyzed (Participants) | 6
    Phase 1: <=18 years | 0
    Phase 1: Between 18 and 65 years | 4
    Phase 1: >=65 years | 2
    Phase 2: number analyzed (Participants) | 19
    Phase 2: <=18 years | 0
    Phase 2: Between 18 and 65 years | 16
    Phase 2: >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 6 Phase 1 patients and 19 Phase 2 patients.
  Participants
    Phase 1: number analyzed (Participants) | 6
    Phase 1: Female | 2
    Phase 1: Male | 4
    Phase 2: number analyzed (Participants) | 19
    Phase 2: Female | 9
    Phase 2: Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were 6 Phase 1 patients and 19 Phase 2 patients.
  Participants
    Phase 1: number analyzed (Participants) | 6
    Phase 1: Hispanic or Latino | 0
    Phase 1: Not Hispanic or Latino | 6
    Phase 1: Unknown or Not Reported | 0
    Phase 2: number analyzed (Participants) | 19
    Phase 2: Hispanic or Latino | 2
    Phase 2: Not Hispanic or Latino | 15
    Phase 2: Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were 6 Phase 1 patients and 19 Phase 2 patients.
  Participants
    Phase 1: number analyzed (Participants) | 6
    Phase 1: American Indian or Alaska Native | 0
    Phase 1: Asian | 0
    Phase 1: Native Hawaiian or Other Pacific Islander | 0
    Phase 1: Black or African American | 0
    Phase 1: White | 6
    Phase 1: More than one race | 0
    Phase 1: Unknown or Not Reported | 0
    Phase 2: number analyzed (Participants) | 19
    Phase 2: American Indian or Alaska Native | 0
    Phase 2: Asian | 1
    Phase 2: Native Hawaiian or Other Pacific Islander | 0
    Phase 2: Black or African American | 1
    Phase 2: White | 13
    Phase 2: More than one race | 0
    Phase 2: Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients With Treatment-Emergent Adverse Events (Phase 1)
Description: In the Phase 1 portion of the study, safety will be assessed after the inclusion of the first 6 patients, to analyze tolerance and adverse events occurring during this trial and will decide on any action to be taken. Safety will be evaluated according to NCI CTCAE V4 criteria. TEAE's were considered adverse events that occurred within 60 days of treatment initiation. The title of this outcome measure was adjusted when results were entered.
Time Frame: 60 days
Population: Phase 1 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib and AML Induction
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Complete Remission Rate (Phase 2)
Description: In Phase 2, the primary endpoint of complete remission rate will be based on IWG 2003 AML response criteria.
  This construct is an overall response composite and it will be assessed using the following metrics:
  Morphologic complete remission (CR): ANC ≥ 1,000/mcl, platelet count ≥ 100,000/mcl, < 5% bone marrow blasts, no Auer rods, no evidence of extramedullary disease. (No requirements for marrow cellularity, hemoglobin concentration).
  Morphologic complete remission with incomplete blood count recovery (CRi): Same as CR but ANC may be < 1,000/mcl but >500 mcl and/or platelet count < 100,000/mcl but >20,000/mcl
  Partial remission (PR): ANC ≥ 1,000/mcl, platelet count > 100,000/mcl, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts < 5% with persistent Auer rods.
  Marrow Leukemia Free State: < 5% bone marrow blasts, no Auer rods, no extra medullary disease. No requirement on cytopenias.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib and AML Induction
Number analyzed (Participants) | 19
Participants
  Complete Remission | 5
  Complete Remission with incomplete counts recovery | 4
  Non-evaluable | 1
  Partial Remission | 1
  Stable Disease | 7
  Progressive Disease | 1

3. Secondary Outcome: Incidence of Hematological Improvement (Phase 2)
Description: Evaluation of hematological improvement will be assessed based on IWG MDS 2006 criteria. Due to differing pretreatment conditions of participants, response to treatment in this construct will be assessed in the following manner:
  Erythroid response (pretreatment <11 g/dL) : Hgb increase at least by 1.5 g/dL. Relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 wk compared with the pretreatment transfusion number in the previous 8 wk. Only RBC transfusions given for a Hgb of below or equal to 9.0 g/dL pretreatment will count in the RBC transfusion response evaluation.
  Platelet response (pretreatment 100x109/L): Absolute increase of at least 30x109/L for patients starting with more than 20x109/L platelets. Increase from less than 20x109/L to more than 20x109/L and by at least 100%.
  Neutrophil response (pretreatment, <1.0x109/L) At least 100% increase and an absolute increase of at least 0.5x109/L.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib and AML Induction
Number analyzed (Participants) | 19
Participants
  Hematological Improvement Erythroid: Yes | 3
  Hematological Improvement Erythroid: No | 13
  Hematological Improvement Erythroid: Missing | 3
  Hematological Improvement Neutrophils: Yes | 6
  Hematological Improvement Neutrophils: No | 10
  Hematological Improvement Neutrophils: Missing | 3
  Hematological Improvement Platelet: Yes | 6
  Hematological Improvement Platelet: No | 10
  Hematological Improvement Platelet: Missing | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for up to 60 days for Phase 1, up to 2 years for Phase 2
Groups:
- Nintedanib and AML Induction: Phase 1; Nintedanib and AML Induction: Phase 2: The AML induction regimen combines Idarubicin 12mg/m2/d day 1 to 3 and Cytarabine 0.667g/m2/d CIV day 1 to 3. Based on the phase I dose, in the randomized phase II, the combination will be compared with chemotherapy+placebo. Nintedanib or placebo will be added at day 8 and continued until end of cycle .
  Nintedanib and AML induction: The AML induction regimen combines Idarubicin 12mg/m2/d day 1 to 3 and Cytarabine 0.667g/m2/d CIV day 1 to 3. In the phase I part, all patients will receive the combination with Nintedanib 200mg bid begun at day 8 and continued until end of cycle. If a significant incidence of dose limiting toxicities is demonstrated, Nintedanib will be given at a lower dose level (150mg bid).
Arm/Group | Nintedanib and AML Induction: Phase 1 | Nintedanib and AML Induction: Phase 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/6 | 8/19
Other Adverse Events (participants affected / at risk) | 6/6 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nintedanib and AML Induction: Phase 1 (N=6) | Nintedanib and AML Induction: Phase 2 (N=19)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cellulitis
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (2) — Oral Abscess
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nintedanib and AML Induction: Phase 1 (N=6) | Nintedanib and AML Induction: Phase 2 (N=19)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 7 (24)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 13 (27)
Nausea (Gastrointestinal disorders) | 3 (3) | 12 (20)
Fatigue (General disorders) | 2 (2) | 6 (8)
Infusion related reaction (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 1 (1) | 7 (10)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 10 (39)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 10 (24)
Blood bilirubin increased (Investigations) | 2 (5) | 6 (15)
Fibrinogen decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 7 (23)
Platelet count decreased (Investigations) | 2 (10) | 6 (39)
White blood cell decreased (Investigations) | 3 (7) | 13 (51)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 11 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 12 (32)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 7 (14)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 5 (7)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (2) | 6 (13)
Insomnia (Psychiatric disorders) | 1 (1) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (9)
Hypertension (Vascular disorders) | 2 (2) | 10 (32)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 6 (8)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Eye disorders - Other (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 8 (13)
Cecal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 9 (15)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (17)
Chills (General disorders) | 0 (0) | 6 (10)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 7 (9)
Fever (General disorders) | 0 (0) | 11 (27)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 1 (1)
Neck edema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 8 (11)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 4 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 9 (16)
Cardiac troponin T increased (Investigations) | 0 (0) | 2 (2)
CPK increased (Investigations) | 0 (0) | 1 (3)
Creatinine increased (Investigations) | 0 (0) | 1 (3)
INR increased (Investigations) | 0 (0) | 7 (8)
Lymphocyte count decreased (Investigations) | 0 (0) | 13 (65)
Weight gain (Investigations) | 0 (0) | 3 (6)
Weight loss (Investigations) | 0 (0) | 3 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 6 (9)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 12 (26)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 8 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 7 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 7 (11)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Othe4 (Nervous system disorders) | 0 (0) | 4 (6)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 3 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 6 (6)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (7)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 4 (8)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT02665143/Prot_SAP_000.pdf